CLINICAL TRIAL: NCT05883163
Title: STIMIT Activator 1 Pivotal Study
Brief Title: STIMIT Activator 1 IDE Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stimit AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-26606
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Diaphragm Issues
Keywords: Non-Invasive Phrenic Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, 1:1 randomized, controlled study using adaptive design
Who Masked: Outcomes Assessor
Masking Description: An independent, blinded Core Lab will analyze the primary endpoint data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Stimulation Group (Experimental): The intervention group will receive non-invasive stimulation of the phrenic nerve for activation of the diaphragm.
  Interventions: Device: Stimit Activator 1
- Control Group (No Intervention): The control group will not received intervention and will be treated with standard of care.

INTERVENTIONS:
Device: Stimit Activator 1 — The Stimit Activator 1 System will be used to stimulate the phrenic nerve resulting in diaphragm activation.
  Arms: Stimulation Group

SUMMARY:
The study is a prospective, multi-center, randomized, controlled study using adaptive design to assess the evidence of safety and performance of the STIMIT Activator 1 System in the treatment of patients who have been mechanically ventilated for up to 7 days and are predicted to require additional minimum 48 hours of mechanical ventilation or longer.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to evaluate the safety and effectiness of the STIMIT Activator 1 System in patients who are on invasive mechanical ventilation (MV) and thus are at risk of diaphragmatic dysfunction/atrophy.

The study is expected to enroll 40 participants at up to 8 centers focusing on North American sites (main focus USA, > 50% of study enrollment from US site). An interim analysis will be conducted after 30 participants have been enrolled and compelted their study follow-up to reconfirm sample size (adaptive design). Participants will be followed for up to 10 days or until they are successfully extubated (weaned) from mechanical ventilation, expire prior to extubation, or withdraw consent.

ELIGIBILITY:
Inclusion Criteria:

1. Are 21 years or older, and,
2. Have recently been placed on invasive MV (enroll and randomized as soon as possible after intubation), and have received no more than 7 days of MV
3. Are predicted to remain on mechanical ventilation for an additional 48 hours or longer post randomization

Exclusion Criteria:

1. Patients that are actively treated with continuous infusion of neuromuscular blocking agents beyond the enrollment period.
2. Medical condition known to affect the phrenic nerve or respiratory muscles (examples of possible medical conditions that could affect the phrenic nerve provided in Annex 1 below).
3. Any patients with ICP probe.
4. Patients with metallic device implants or body penetrating metallic devices in the upper body area within 30cm (12inches) from the coils; known anatomy or devices in the neck area (e.g., ECMO cannulas in the neck area, collars or cranial appliances) that would interfere with headset placement or stimulation.
5. Any non-removable electrical / electronic device (device internal or external) that may be prone to interaction with, or interference from the STIMIT Activator, such as pacemakers, implantable defibrillators, implanted medication pumps, bio-stimulators, deep brain stimulators, implanted nerve stimulator, deep brain stimulators or cochlear device implants.
6. BMI >40.
7. Cardiogenic or septic shock with ongoing severe hemodynamic instability that cannot be stabilized within the enrollment period.
8. Physician thinks that the patient will not tolerate initial installation of the STIMIT respiratory sensor.
9. Anticipating withdrawal of life support and/or shift to palliation as the goal of care.
10. Known to be pregnant.
11. Participating in another clinical trial studying an experimental Intervention that could affect the study primary outcome.
12. Patients whose ultrasonographic assessment of right-sided diaphragmatic thickness would be too difficult (e.g. local subcutaneous emphysema surrounding the zone of apposition, large dressings in the zone of apposition that cannot be removed).
13. Patients with neck condition that would not allow placing the coils on the neck (e.g. open wounds that cannot be covered, skin at risk for burns).
14. Patients with significant spontaneous efforts (P0.1 < - 2) that would not be at risk for diaphragmatic atrophy/ dysfunction.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Efffectiveness: Preservation of Diaphragm Thickness | Up to Day 10
  The intra-individual change in diaphragm thickness will be measured daily via ultrasound and compared between intervention and control groups.
Safety: Rate of device or procedure related serious adverse events (SAEs) | Up to Day 10
  Events will be collected for intervention group during the course of treatment.

SECONDARY OUTCOMES:
Preservation of Diaphragm Thickness | Up to Day 3
  The intra-individual change in diaphragm thickness will be measured daily via ultrasound and compared between intervention and control groups.
Time to Rapid Shallow Breathing Index (RSBI) < 105 | Up to Day 10
  Time from intubation to RSBI<105 breaths/min/L in days will be compared between intervention and control groups.
Maximum Inspiratory Pressure (MIP) at extubation | Up to Day 10
  MIP at extubation will be compared between intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, MD, Principal Investigator — St Michael's Hospital Unity Health Toronto
Locations (4):
- United States (3):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Virginia Medical Center, Charlottesville, Virginia
- St Michael's Hospital Unity Health Toronto, Toronto, Canada

REFERENCES:
- [Derived] Schreiber AF, Subira C, Sklar M, Santos M, Ko M, Panelli A, Schaller SJ, Theodore D, Rowley DD, Watson D, Bonde P, Baedorf Kassis EN, Talmor DS, Ranieri M, Goligher EC, Slutsky A, Brochard LJ. Multi-center randomized superiority clinical trial in the early phase of mechanically ventilated patients to preserve diaphragm thickness using non-invasive magnetic phrenic nerve stimulation: STIMIT ACTIVATOR 1 pivotal trial. Trials. 2025 Jun 11;26(1):202. doi: 10.1186/s13063-025-08838-2. PMID 40500715